CLINICAL TRIAL: NCT03889899
Title: A Safety and Effectiveness Study of Intratumoral Diffusing Alpha Radiation Emitters for the Treatment of Malignant Cutaneous, Mucosal or Superficial Soft Tissue Neoplasia
Brief Title: Alpha Radiation Emitters Device (DaRT) for the Treatment of Cutaneous, Mucosal or Superficial Soft Tissue Neoplasia.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Alpha Tau Medical LTD. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CTP-CMN-03
Record Dates: First submitted 2019-03-21; First posted 2019-03-26 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Skin Cancer; Mucosal Neoplasm of Oral Cavity; Soft Tissue Neoplasm
Keywords: Squamous Cell Carcinoma; SCC; Skin Cancer; Skin metastasis; HNSCC; Carcinoma, Squamous; CMN; Basal cell carcinoma; Superficial sarcoma; Kaposi sarcoma; Alpha radiation; Cutaneous lesion; Tongue cancer; Lip cancer
MeSH Terms: conditions — Skin Neoplasms; Soft Tissue Neoplasms; Carcinoma, Squamous Cell; Squamous Cell Carcinoma of Head and Neck; Carcinoma, Basal Cell; Sarcoma, Kaposi; Tongue Neoplasms; Lip Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- DaRT Seeds (Experimental): Intratumoral Diffusing alpha-emitters Radiation Therapy (DaRT) Seeds
  Interventions: Device: Radiation: Diffusing Alpha Radiation Emitters Therapy (DaRT)

INTERVENTIONS:
Device: Radiation: Diffusing Alpha Radiation Emitters Therapy (DaRT) — An intratumoral insertion of a seed(s), loaded with Radium-224, securely fixed in the seeds. The seeds release by recoil into the tumor short-lived alpha-emitting atoms.

SUMMARY:
A unique approach for cancer treatment employing intratumoral diffusing alpha radiation emitter device for superficial cutaneous, mucosal or soft tissue neoplasia

DETAILED DESCRIPTION:
This will be a prospective, open label, single arm, controlled study, assessing the safety and efficacy of diffusing alpha emitters radiation therapy (DaRT) delivered through radioactive seeds inserted into the tumor.

This approach combines the advantages of local intratumoral irradiation of the tumor, as used in conventional brachytherapy, with the power of the alpha radiation emitting atoms, that will be introduced in quantities considerably lower than radiation therapy already used in patients.

Superficial lesions with histopathological confirmation of malignancy will be treated using DaRT seeds.

Reduction in tumor size 70 days after DaRT insertion will be assessed. Safety will be assessed by the incidence, severity and frequency of all Adverse Events (AE).

ELIGIBILITY:
Inclusion Criteria:

* Subjects with histopathological confirmation of primary or secondary malignant cutaneous neoplastic lesions, or oral cavity mucosal tumors, or superficial soft tissue sarcoma.
* Subjects with a tumor size ≤ 7 centimeters in the longest diameter.
* Measurable disease according to RECIST v1.1.
* Subjects over 18 years old.
* Subjects' ECOG Performance Status Scale is < 2.
* Subjects' life expectancy is more than 6 months.
* Platelet count ≥100,000/mm3.
* International normalized ratio of prothrombin time ≤1.8.
* Creatinine ≤1.9 mg/dL.
* Women of childbearing potential (WOCBP) will have evidence of negative pregnancy test.
* Subjects are willing to sign an informed consent form.

Exclusion Criteria:

* Subject has a tumor of Keratoacanthoma histology.
* Patients with significant comorbidities that the treating physician deems may conflict with the endpoints of the study (e.g., poorly controlled autoimmune diseases, vasculitis, etc.)
* Patients undergoing systemic immunosuppressive therapy excepting intermittent, brief use of systemic corticosteroids
* Volunteers participating in another interventional study in the past 30 days which might conflict with the endpoints of this study or the evaluation of response or toxicity of DaRT.
* High probability of protocol non-compliance (in opinion of investigator).
* Subjects not willing to sign an informed consent.
* Women who are pregnant or breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-10-21 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Tumor response to DaRT | 9-11 weeks after DaRT seed insertion.
  Assessment of the rate of malignant cutaneous, mucosal or superficial soft tissue tumors response using the Response Evaluation Criteria in Solid Tumors (RECIST) (Version 1.1)
Adverse Events | Time Frame: 9-11 weeks post DaRT insertion.
  The incidence, frequency, severity and causality of acute adverse events related to the DaRT treatment

SECONDARY OUTCOMES:
Assessment of the reduction in tumor volume | 9-11 weeks follow-up visit.
  Assessment of the reduction in tumor volume based on CT / PET-CT measured tumor volume
DaRT seeds placement. | Day of insertion procedure.
  Assessment of the DaRT seeds placement by localization of the DaRT seeds in the tumor using CT imaging on the day of DaRT insertion.
Change in quality of life | Screening, DaRT removal and day 70 visits.
  Assessment of patient reported health-related Quality of Life outcome after DaRT, using QoL questionnaire Skindex-16 questionnaire score. An overall score ranging from 0 (best) to 100 (worst).
Change in quality of life | Screening, DaRT removal and day 70 visits.
  Assessment of patient reported health-related Quality of Life outcome after DaRT, using QoL questionnaire Skin Cancer Index (SCI) questionnaire score. An overall score ranging from 0 (best) to 100 (worst).

CONTACTS AND LOCATIONS:
Overall Officials: Tomer Charas, MD, Principal Investigator — Radiotherapy unit at Rambam Health Care Campus, Israel
Locations (1):
- RAMBAM Health Care Campus, Haifa, Israel

IPD SHARING:
Plan to Share IPD: No